CLINICAL TRIAL: NCT02479178
Title: A Phase 2 Study to Determine the Efficacy and Safety of BIND-014 (Docetaxel Nanoparticles for Injectable Suspension) in Patients With Urothelial Carcinoma, Cholangiocarcinoma, Cervical Cancer and Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Study of BIND-014 in Patients With Urothelial Carcinoma, Cholangiocarcinoma, Cervical Cancer and Squamous Cell Carcinoma of the Head and Neck
Acronym: iNSITE2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: BIND Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIND-014-008
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Urothelial Carcinoma; Cholangiocarcinoma; Cervical Cancer; Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Carcinoma, Transitional Cell; Cholangiocarcinoma; Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck

INTERVENTIONS:
Drug: BIND-014 (docetaxel nanoparticles for injectable suspension) — docetaxel nanoparticles for injectable suspension

SUMMARY:
BIND-014 (docetaxel nanoparticles for injectable suspension) is being studied in patients with advanced urothelial carcinoma, cervical cancer, cholangiocarcinoma or carcinomas of the biliary tree and squamous cell carcinoma of the head and neck.

Ferumoxytol imaging will also be investigated at US sites as an exploratory endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced urothelial carcinoma, cervical cancer, cholangiocarcinoma or carcinomas of the biliary tree or squamous cell carcinoma of the head and neck.
2. Progressive disease after ≥ 1 prior chemotherapy regimen.
3. Patients with brain metastases are eligible if asymptomatic and neurologically stable for at least 4 weeks and are not taking any medications contraindicated
4. Chemotherapy must have been completed at least 4 weeks prior to initiation of study medication
5. ECOG performance status 0-1
6. Tumors must have measurable disease as per RECIST (version 1.1);
7. Female or male, 18 years of age or older
8. Adequate organ function
9. Life expectancy of > 3 months

Exclusion Criteria:

1. Current treatment on another therapeutic clinical trial
2. Prior treatment with docetaxel within 6 months of enrollment
3. Stage II, III or IV cardiac failure
4. Carcinomatous meningitis
5. Ongoing cardiac dysrhythmias
6. Peripheral neuropathy
7. Serious concomitant conditions
8. Pregnant or breast feeding
9. Known sensitivity to ferumoxytol
10. Hypersensitivity to polysorbate 80

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
To determine the objective response rate (ORR) in patients with advanced urothelial carcinoma (transitional cell carcinoma), cervical cancer, cholangiocarcinoma or carcinomas of the biliary tree and squamous cell carcinoma of the head and neck. | 18 weeks
  Patients will be followed for ORR for an expected average of 18 weeks

SECONDARY OUTCOMES:
Progression Free Survival | Change in tumor size will be assessed using RECIST measurements. RECIST assessments will be carried out at baseline, week 6, week 12 and every 6 weeks thereafter relative to first dose of study drug, an expected average of 18 weeks.
Overall Survival | Participants will be followed for survival, an expected average 24 weeks after treatment discontinuation
Best Response | Change in tumor size will be assessed using RECIST measurements. RECIST assessments to be carried out at baseline, week 6, week 12 and every 6 weeks thereafter relative to first dose of study drug, an expected average 18 weeks
Duration of Response | Change in tumor size will be assessed using RECIST measurements. RECIST assessments to be carried out at baseline, week 6, week 12 and every 6 weeks thereafter relative to first dose of study drug, an expected average 18 weeks
Time to Response | change in tumor size will be assessed using RECIST measurements. RECIST assessments to be carried out at baseline, week 6, week 12 relative to first dose of study drug
Disease Control Rate | Change in tumor size will be assessed using RECIST measurements. RECIST assessments to be carried out at baseline, week 6, week 12 and every 6 weeks thereafter relative to first dose of study drug, an expected average 18 weeks
Safety and Tolerability, as measured by number of participants with adverse events | Measured from first dose of study drug until 30 days after study discontinuation

CONTACTS AND LOCATIONS:
Locations (23):
- United States (8):
  - Investigative Site: #20, Goodyear, Arizona
  - Investigative Site: #42, Greenbrae, California
  - Investigative Site: #39, Denver, Colorado
  - Investigative Site: #34, Detroit, Michigan
  - Investigative Site: #34, St Louis, Missouri
  - Investigative Site: #43, Las Vegas, Nevada
  - Investigative Site: # 37, Oklahoma City, Oklahoma
  - Investigative Site: # 33, San Antonio, Texas
- Russia (15):
  - Investigative Site: #74, Arkhangelsk
  - Investigative Site: #75, Kazan'
  - Investigative Site: #70, Moscow
  - Investigative Site: #80, Murmansk
  - Investigative Site: #81, Omsk
  - Investigative Site: #84, Saint Petersburg
  - Investigative Site: #85, Saint Petersburg
  - Investigative Site: #73, Saint Petersburg
  - Investigative Site: #78, Saint Petersburg
  - Investigative Site: #79, Saint Petersburg
  - Investigative Site: #88, Saratov
  - Investigative Site: #77, Sochi
  - Investigative Site: #72, Ufa
  - Investigative Site: #87, Ulyanovsk
  - Investigative Site: #82, Yaroslavl